CLINICAL TRIAL: NCT02733809
Title: Mechanism of Sorafenib Resistance in Patients With Advanced Hepatocellular Carcinoma
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Saud University (Other)
Collaborators: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Principal Investigator, Mazen Hassanain, Assocaite Professor of Surgery and Consultant HPB and Transplant Surgery, King Saud University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: KSULDRCSSMH001
Record Dates: First submitted 2016-02-15; First posted 2016-04-12 (Estimated); Last update posted 2019-08-20 (Actual); Status verified 2019-08

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Sorafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sorafenib (Experimental): Group under the treatment ( sorafenib ) Maximum dose of 400 mg BID If subjects devolves adverse events, dose can be reduced.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — Liver lesion biopsy (HCC) and blood samples will be taken from the subjects before starting the treatment course, and another biopsy and blood samples when they devolve a resistance.
  Other Names: Nexavar

SUMMARY:
It has been shown previously that gene expression profiling signature (a set of dysregulated genes) can be used for molecular classification, diagnosis, and prognosis of several types of cancers. In This study the hypothesise that resistant tumor may be due to genetic mutations and/or other alternative pathways that could be the reason to overcome the Sorafenib and still proliferate.

Primary objectives To evaluate the primary and secondary potential mechanisms by which HCC patients on Sorafenib treatment would be resistant to therapy and also identify the favorable genetic makeup of patients responding to treatment.

Measures of primary outcome:

* cDNA microarray analysis on the MAP kinase pathway.
* mRNA quantification of genetic expression (RT-PCR) for identification of upregulated genes, and confirmed by corresponding proteomic testing (by Mass Spectroscopy) in the serum for potential serum markers. Secondary Objectives Progression free survival: Time to disease progression in patients in Saudi Arabia with HCC receiving Sorafenib: [defined as time, in weeks, from the baseline visit to progression of the disease or death from any cause] will be diagnosed using the RECIST criteria based on a trimestrial abdominal CT evaluation.
* Survival rates and Predictors of survival:

  * Survival defined as the time from baseline visit to death from any cause [in weeks].
  * Variables identified in multivariate regression analysis from overall treated patients independently associated with survival till study completion or death. Justification and Value to the Kingdom Sorafenib in the treatment of advanced HCC is a recent development. Since the only current effective treatment for advanced HCC is resection or transplantation and the list for these procedures are ever-growing due to the confounding effect of the lack of infrastructure in the Kingdom, selecting treatment for patients who are more likely to respond to Sorafenib treatment The Long-Term Comprehensive National Plan for Science, Technology and Innovation will help to reduce costs of managing HCC. Among Saudi Arabia population, there are a unique set of patients here (e.g. non-alcohol related HCC, genotype 4 HCV patients and genotype D HBV patients, high percentage of obese patients i.e. NASH) which is different from other parts of the world. There is increasing incidence of HCC in Saudi Arabia. Due to available expertise in management of HCC patients in the participating institutions in the study, this project will represent a bridge for the transfer of technology so that our research staff and doctors will have more expertise in carrying out these techniques independently. This study will also run in parallel to the on-going initiative to start a HCC biobanking establishment which will provide the samples needed to carry out our genetic studies in future. Finally, since the use of Sorafenib (at present, the only approved treatment for advanced HCC) in the treatment of advanced HCC is a new field, the findings of our study will have important implications in the management of HCC, both locally and internationally.

HCC is the third most common cancer in Saudi Arabia. In 2001, HCC was the second most common cancer affecting Saudi males and the eighth most common cancer affecting females. Most of patients (90%) present at a more advanced stage when symptoms prevail.

Given the high prevalence of HCC in the Kingdom, it is pertinent to study why some patients are resistant to Sorafenib compared to others. Elucidation of the differences in mechanisms among responders and non-responders to Sorafenib therapy will enable physicians to make better decisions in terms of treating Saudi HCC patients.

DETAILED DESCRIPTION:
Introduction Hepatocellular carcinoma (HCC) is a major health problem, accounting for more than 626,000 new cases per year worldwide. It is the third highest cause of cancer-related death globally. In the west, the disease is diagnosed in 30 to 40% of all patients at early stages and is amenable to potentially curative treatments, such as surgical therapies (resection and liver transplantation) and locoregional procedures (radio-frequency ablation). There are no clear epidemiological studies in the Kingdom of Saudi Arabia that gives the real incidence of HCC in Saudi population, however the Saudi Cancer registration have labelled it as among the top five cancers in the country. Sorafenib has emerged as the treatment of choice in the treatment of advanced HCC and has demonstrated an anti-angiogenic and anti-proliferative effect. It is a kinase inhibitor that decreases tumor cell proliferation in Vitro. Sorafenib has been shown to inhibit multiple intracellular (CRAF, BRAF, and mutant BRAF) and cell surface kinases (KIT, FLT-3, RET, VEGFR-1, VEGFR-2, VEGFR-3 and PDGFR-B). Several of these kinases are thought to be involved in tumor cell signaling, angiogenesis and apoptosis. In a phase 3 international, multi-center, randomised, doubleblind, placebo-controlled trial in patients with unresectable hepatocellualr carcinoma Sorafenib showed a statistically significant advantage over placebo for overall survival (HR: 0.69, p=0.00058). Final analysis of time to tumor progression also was significantly longer in the Protocol number: 1.0 dated 01Aug2013 Short title: HCC - Sorafenib study Confidential Page 11 The Long-Term Comprehensive National Plan for Science, Technology and Innovation Sorafenib arm. This benefit was calculated in months because of the quick emergence of resistance in many patients. Therefore, individualizing the treatment to patients with most expected response and avoiding it in patients with resistant cancers has stimulated this research to evaluate why some patients develop resistance to this therapy.

Literature review Epidemiology Hepatocellular carcinoma (HCC) is the sixth most common cause of cancer worldwide with an annual incidence of over 711,000 new cases, and the third most common cause of cancer death with an annual mortality of 679,000 patients. Most commonly HCC develops in cirrhosis, irrespective of the etiology. In the western world, chronic alcohol abuse and nonalcoholic stratohepatitis are about the as important etiologic factors for cirrhosis as chronic hepatitis c. In chronic hepatitis C it is estimated that about 20% of patients will eventually develop cirrhosis after 20-30 years of infection. Once cirrhosis is established, the annual risk of developing HCC is estimated to be between 3 and 4 %, largely irrespective of the etiology of cirrhosis. Diagnosis of HCC HCC is mostly asymptomatic in early stage disease. Without proper surveillance programs of cirrhotic patients, diagnosis is only established in advanced stage disease. The efficacy of surveillance by Ultrasound (and to a lesser extent by alpha-fetoprotein measurement) has been established in prospective trials in the west as well in the east. surveillance by experienced sonographers makes curative treatment possible treatment possible in up to 75% of patients,while there is no curative treatment without proper surveillance. Surveillance is recommended for the following groups of patients: Hepatitis B carriers Asian males > 40 years, Asian females >50 years, All cirrhotic hepatitis B carriers, Family history of HCC, Africans over age 20. For non-cirrhotic hepatitis B carriers not listed above the risk of HCC varies depending on the severity of the underlying liver disease, the Long-Term Comprehensive National Plan for Science, Technology and Innovation inflammatory activity. Patients with high HBV DNA concentrations and those with ongoing hepatic inflammatory activity remain at risk for HCC. Non-hepatitis B cirrhosis Hepatitis C, Alcoholic cirrhosis, Genetic hemochromatosis, Primary biliary cirrhosis. Although the following groups have an increased risk of HCC no recommendations for or against surveillance can be made because a lack of data precludes an assessment of whether surveillance would be beneficial - Alpha1-antitrypsin deficiency ,Non-alcoholic steatohepatitis, Autoimmune hepatitis. Once a lesion is detected by ultrasound, the diagnosis can be established radiologically in lesions with typical appearance above 1 cm in diameter. Biopsy is mandated only in cases with atypical presentation on imaging. Staging of HCC Staging of HCC can be done using several systems. currently, the most widely used staging system is the Barcelona Clinic Liver Cancer (BCLC) staging system , which takes the underlying liver disease, tumor characteristics, as well as the general performance status into account . This staging system is popular as it is directly linked to treatment, making treatment decisions easy. Advanced stage HCC: the current role of medical therapies In western countries, about 30 % of patients are identified with an HCC in BCLC stage 0 or A, either through surveillance or by chance. For those patients curative options can be applied, which currently involve only surgical or interventional treatments. However , curatively treated patients , except for those who underwent transplantation, will have a tumor recurrence in 70 to 80 % of cases within 5 years of therapy and will eventually progress to BCLC B or BCLC C stage disease. Another 20 % of patients are diagnosed at very advanced stages BCLC D, being either symptomatic from the decompensated cirrhosis (Child-Pugh C) or having an advanced tumor. Those patients have a very short survival, which cannot be influenced by any therapeutic intervention and are only eligible to receive best supportive care. Currently, the domain of medical therapies for HCC is in the setting of advanced stage BCLC C. Conventional chemotherapy of any kind has never shown any meaningful therapeutic benefit, particularly in overall survival in randomized controlled trials in adult patients and cannot be recommended for the treatment of HCC today. Conventional cisplatin-based chemotherapy, Technology and Innovation without doxorubicine only has a place in the treatment of childhood hepatoblastoma, which is a distinctly different disease entity. In hepatoblastoma cisplatin-based chemotherapy does improve survival and can even provide a cure in over 80% of patients when combined with resection. Medical treatment of HCC changed dramatically in 2007 , when the first data from the successful use of targeted agents in advanced stage HCC, in particular tyrosine kinase inhibitors, were presented. Up-regulated signaling through the mitogen-activated protein kinase (MAPK) intracellular signal transduction pathway plays a crucial role in the development of hepatocellular carcinoma , as does tumor angiogenesis .The MAPK pathway comprises Raf ,MAPK kinase (MEK ) and extracellular signal-regulated Kinase (ERK), and is a mediator of tumor proliferation, differentiation and survival. The identification of pivotal pathways, such as the MAPK cascade, led to the development of targeted treatments, such as Sorafenib. Sorafenib is an orally active multikinase inhibitor that inhibits cell surface tyrosine kinases, as well as downstream intracellular Raf kinases in the MAPK cascade. Sorafenib is widely available for the use in the treatment of advanced renal cell carcinoma and has been reviewed in this indication previously. Recently, Sorafenib was also approved in the US and the EU for use in the treatment of hepatocellular carcinoma, the first systemic drug to be approved in this indication. Indeed, current US treatment guidelines recommend Sorafenib as the first-lone treatment option in patients with unresectable HCC who are Child-Pugh class A. Receptor tyrosine Kinases inhibited by Sorafenib include vascular endothelial growth factor receptor (VEGFR)-1, VEGFR-2, VEGFR-3, Platelet-derived growth factor receptor (PDGFR)-B, cKIT, FMS-like tyrosine kinase 3 (FLT-3) and RET. Intracellular Raf serine/threonine kinase isoforms inhibited by Sorafenib include Raf-1(or C-Raf), wild -type B-Raf and Mutant B-Raf. These kinases are involved in tumor cell proliferation and tumor angiogenesis. In vitro, dose-dependent inhibition of cell proliferation was seen with Sorafenib in the human hepatocellular carcinoma cell lines PLC/PRF/5 and HepG2. Moreover, dose dependent induction of apoptosis was seen after Sorafenib exposure, as assessed by TUNEL (terminal deoxynucleotide transferase d-uridine triphosphate nick end labeling) staining. Inhibition by Sorafenib of the Raf/MEK/ERK signaling pathway in PCL/PRF/5 and HepG2 cells was shown by, among other things, the inhibition of MEK and ERK phosphorylation. Sorafenib demonstrated Protocol number: 1.0 dated 01Aug2013 Short title: HCC - Sorafenib study Confidential Page 14 The Long-Term Comprehensive National Plan for Science, Technology and Innovation dose-dependent antitumor activity in murine xenograft model of PCL/PRF/5 human hepatocellular carcinoma. Significant tumor growth inhibition of 49% and 78% was seen in mice receiving oral Sorafenib 10 or 30 mg/kg/day for 16 or 21 days ( both P 16 weeks and 48 (35.0%) had progressive disease (the remaining 32 patients [23.4%] were not available for independent review). With Sorafenib, the median time to progression was 4.2 months (investigator assessment) or 5.5 months (independent assessment), and the median overall survival duration was 9.2 months. Phase III trial The clinical efficacy of oral Sorafenib was examined in patients with advanced HCC in a randomized, double-blind, placebo-controlled, multi center, phase III trial (the SHARP study) (22). Inclusion criteria were histologically proven, advanced hepatocellular carcinoma, with at least one measurable untreated lesion, an ECOG performance status of 0-2, Child-Pugh class A and no prior systemic treatment . 902 patients were screened and 602 were randomized to receive oral Sorafenib 400 mg twice daily (n=299) or placebo (n=303). The median duration of treatment was 23 weeks in Sorafenib recipients and 19 weeks in placebo recipients. Prior to randomization, patients were stratified according to macroscopic vascular invasion and/or extrahepatic spread, ECOG performance status and Geographical region. In terms of baseline characteristics, mean patient age was 65.5 years; 87% of patients were male; 87.5% of patients were from Europe; 96.5% of patients were Child-Pugh class A; 54%, 38.5% and 7.5% of patients had an ECOG performance status of 0, 1, 2 at baseline; 17.5% and 82.5% of patients had Barcelona Clinic Liver Cancer Group stage B and C cancer; and 70% of patients had vascular invasion and/or extrahepatic spread . The primary endpoints were overall survival and time to symptomatic progression (defined as the time from randomization to a 4-point decline from baseline in patient response to the Functional Assessment Of Cancer Treatment Hepatobiliary Symptom index [FHSI-8] confirmed at next visit , deterioration to ECOG performance status 4, or death). The time to progression (assessed by independent central review) was a pre-specified secondary endpoint. Tumor response rates were assessed using Response Evaluation Criteria in Solid Tumors (RECIST). Analyses were conducted in the intent-to-treat (ITT) population (22). Sorafenib significantly improved survival in patients with advanced hepatocellular carcinoma in the SHARP trial (22). The median duration of survival was 10.7 months with Sorafenib and 7.9 months with placebo, yielding a hazard ratio (HR) of 0.69 (95% CI 0.55, 0.88; P = 0.00058). Following the second planned interim analysis, the SHARP study was terminated early on the basis of this survival result. At the time of study termination, there was no significant difference between Sorafenib and placebo recipients in the time to symptomatic progression (assessed using FHSI-8 criteria). The median time to progression (assessed by independent central review) was significantly longer in patients receiving Sorafenib than those receiving placebo (5.5 vs. 2.8 months), with an HR of 0.58(95% CI 0.44, 0.74; P Overall study design Screening and Pre-Treatment Period Investigator/ Co-Investigator/Study Coordinator • Medical history • Biopsy and review of pathology • Physical examination and vital signs • Review of previous or concurrent medications and procedures • Child-Pugh assessment • ECOG assessment • Lesion(s) measurement • Determination of study eligibility • Written, signed and date informed consent Laboratory investigations • Hematology: CBC, Differential • Serology: HBV, HCV, and HIV • The levels of the Bimarkers: c-KIT, Soluble VEGFR-2,-3. • Coagulation: platelets, PT, PTT, INR • Liver function tests • Serum pregnancy test (as appropriate) Radiological investigations • CT scan (or MRI) of the chest • CT scan (or MRI) of the abdomen • PET Scan Patient • Review of patient information leaflet Treatment period Baseline Visit - Day 1 Investigator/ Co-Investigator/Study Coordinator • Review of concomitant medications and therapies • Review of ECOG • Prescription of Sorafenib Patient • Start of the Sorafenib 6-8 weeks cycle Sorafenib Cycle Week 0-6/8 Laboratory investigations to be done on a weekly basis • Hematology: CBC, Differential • Serology: HBV, HCV, and HIV • Coagulation: platelets, PT, PTT, INR results of laboratory investigations on a weekly basis • See patients every other week Patient • Takes the appropriate dose of Sorafenib • Goes for blood test every week • Consult with the investigator/co-investigator every other week Visit after first Sorafenib cycle (Week 5 + 1 week) Investigator/ Co-Investigator/Study Coordinator • Physical examination • Review of concomitant medications and therapies • Child-Pugh re-assessment • ECOG re-assessment • Lesion(s) measurement • Recording of Adverse events Laboratory investigations • Hematology: CBC, Differential • Coagulation: platelets, PT, PTT, INR • Liver function tests Radiological investigations • CT scan (or MRI) of the abdomen Follow-up Visits (Every 3 months)* Investigator/ Co-Investigator/Study Coordinator • Physical examination • Review of concomitant medications and therapies • Child-Pugh re-assessment • ECOG re-assessment • Lesion(s) measurement • Recording of Adverse events Laboratory investigations • Hematology: CBC, Differential • Coagulation: platelets, PT, PTT, INR • The Bio-markers: c-KIT, VEGFR -2,-3 at week 12. • Liver function tests Radiological investigations • CT scan (or MRI) of the abdomen *The patient is going to be followed up in the basis of either stable disease or partial response or progression this based on radiological profession (which is assessed by RECIST). For those with progression other Biopsy will be taken and the tissue to be evaluated further.

Study procedures All laboratory tests will be conducted as normal with additional specific tests to be performed in Liver Disease Research Center (LDRC), or the Proteomics Lab, KSU-Riyadh. Blood will be collected in three 7ml tubes with each biopsy. cDNA microarray analysis will be done on the pathways acted on by Sorafenib, namely the MAP kinase pathway. The analysis will be done at LDRC, KSU-Riyadh. • Tissue samples will be obtained in all patients from the tumor under imaging guidance • Tumor tissue biopsies will be performed at baseline and at end-of-study/when study endpoint is met o A minimum of 3 cm of tumor tissue will be obtained (2-3 needle passes). o Transportation of samples to the LDRC will be done on dry ice. o Tissue obtained will be snap frozen at -800C until processing. o Tissue will be tested for genes involved in the RAF pathway. o Genetic expression from the fresh tumor tissue will be quantified using RT-PCR for mRNA quantification. Once upregulated genes are identified, their corresponding proteomic expression will be tested in the serum for potential serum markers. Proteomic testing will be performed using Mass Spectroscopy. Additional specific blood tests will be performed in LDRC. Blood will be collected in two 7 ml EDTA tubes (purple top) and one plain tube (red top). Blood samples will be collected at the same time with the liver biopsy. Blood once collected will be transported immediately to LDRC on dry ice and stored at -80oC. Samples will be thawed and data analysed when the individual patient has met study end-point or at study completion, as relevant. Liver biopsy samples will also be transported on dry ice to LDRC and snap-frozen at -80oC for subsequent analysis. Blood and tissue will be collected and transported by pre-arrangement with LDRC staff, and will be coordinated by the SOLID registrar (Nouf Alanezi) and/or the study CRC in KAMC-Riyadh. All patient-related data, including demographic, clinical, laboratory, and radiological data will be collected in the comprehensive HCC eCRF of the SOLID registry where appropriate. As a feature of the registry, all patient-related data is encoded in order to remove any patient identifiers. All blood samples stored for end-of-study investigations will be barcoded and the stickers tagged to the SOLID registry identifiers for easy retrieval.

Study subjects The study is expected to run for about 3 years and patients will be followed for a period of 24 months. All consecutive patients presenting with HCC satisfying study inclusion and exclusion criteria will be approached for participation. At an average, about 200 patients with HCC are evaluated annually in the multi study centres. We anticipate that 60 patients would be eligible for the study of whom 40 would be recruited for the study. A total of 40 patients will be recruited from 2 - 3 centers in KSA (KSU, LDRC; KAMC-Riyadh). Of these 15 patients will be recruited from King Abdulaziz Medical City, Riyadh. Recruitment is planned to be completed in the first year of the study.

Duration of treatment and removal of subjects Patients will be followed for a period of 24 months. Patients removed from study for unacceptable adverse events will be followed until resolution or stabilization of the adverse event. Patients are to continue therapy with Sorafenib until • Disease progression • Until a criterion is met for stopping therapy like o Concurrent illness that prevents further administration of treatment o Unacceptable adverse events(s) o Patient decides to withdraw from the study o General or specific changes in the patient's condition render the patient unacceptable for further treatment in the judgment of the investigator. In the event of radiologic progression, patients may continue to receive the study drug. Decisions about continuing study medication will be made at the discretion of the investigator, based on the investigator's judgment about the patient's clinical status. In general, it is suggested that patients remain on Sorafenib if, in the opinion of the investigator, the patient may be benefiting from continuing on study drug Removal of subjects and the reason of the removal will be documented.

Treatment description No investigational or commercial agents or therapies other than Sorafenib may be administered with the intent to treat the patient's malignancy. Sorafenib will be given at the dose of 2 tablets of 200mg (400 mg) to be taken twice a day in the morning and in the evening without food (at least 1 hour before or 2 hours after a meal). If a dose reduction is necessary, the Sorafenib dose may be reduced to 200 mg twice a day. If additional dose reduction is required, the dose may be reduced to a single 400 mg dose every other day. Reported adverse events, potential risks, and appropriate dose modifications for are described below. Informed Consent: If a patient is found to meet the eligibility criteria and expresses an interest in participation, Other treatment options will also be discussed with the patient prior to completing informed consent. No study related procedures will be conducted prior to the patient signing the informed consent. The subject will be provided with a copy of the Patient Information Sheet and will be given the opportunity to ask any question or seek clarification.

ELIGIBILITY:
Inclusion Criteria:

Male or female patient over 18 years of age

* Patient who have a life expectancy of at least 12 weeks
* Biopsy proven diagnosis of hepatocellular carcinoma
* Liver lesions are visible and measurable of at least 3 cm in size
* Advanced HCC, defined by the presence of one of the followings:

  * Vascular invasion
  * HCC with cancer-related symptoms with ECOG Score of 0, 1 or 2
  * Progression after resection or local ablation and not for further curative therapies
* Cirrhotic status of Child-Pugh class A and B (score ≤ 8)
* The following laboratory parameters:

  * Platelet count > 50 X 109 /L
  * Hemoglobin > 85 g/L
  * Total bilirubin < 51.3 umol/L
  * ALT and AST < 5X upper limit of normal
  * Amylase and lipase < 1.5 X the upper limit of normal
  * Serum creatinine < 1.5 X the upper limit of normal
  * Prothrombin time (PT) international normalized ratio (INR) < 2.3 or PT < 6 seconds above control. Patients who are being therapeutically anticoagulated with an agent such as Coumadin or heparin will be allowed to participate provided that no prior evidence of underlying abnormality in these parameters exists.
* Able to give written informed consent prior to any study specific screening procedures with the understanding that the patient has the right to withdraw from the study at any time, without prejudice.
* Any institution/centre specific criteria that must be adhered to for the patient to be eligible.

Exclusion Criteria:

Previous or concurrent cancer that is distinct in primary site or histology from HCC.

Except:

* Cervical carcinoma in situ
* Prostate cancer with good prognosis
* Treated basal cell carcinoma
* Superficial bladder tumors (Ta, Tis & T1)
* Any cancer curatively treated 3 years prior to entry is permitted.

  * A Child-Pugh rating of C at entry
  * An ECOG performance score of 3 or 4 at entry
  * Extensive extra-hepatic disease
  * Tumor volume > 50% of liver volume
  * Contraindication to angiography or selective visceral catheterization
  * Any bleeding diathesis or coagulopathy that is not correctable by usual therapy or hemostatic agent
  * Severe peripheral vascular disease precluding catheterization
  * History of severe allergy or intolerance to contrast agents, narcotics, sedatives or atropine that cannot be managed medically
  * Platelet count < 30,000 or < 50% prothrombin activity
  * Renal failure requiring hemo-or peritoneal dialysis
  * Pulmonary insufficiency (clinically evident history of chronic obstructive pulmonary disease)
  * History of cardiac disease:

    * Congestive heart failure > New York Heart Association (NYHA) class2
    * Active coronary artery disease
    * Uncontrolled hypertension
  * Active clinically serious infection(s)
  * Known history of human immunodeficiency virus (HIV) infection
  * Patient with clinically significant gastrointestinal bleeding within 30 days prior to study entry
  * History of organ allograft/transplantation
  * Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
  * Known or suspected allergy to the investigational agent or any agent given in association with this trial
  * Patients unable to swallow oral medications
  * Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study
  * Pregnant or breast-feeding patients
  * Women of childbearing potential must have a negative pregnancy test performed within seven days prior to the start of study drug.
  * Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial.

Excluded therapies and medications - previous and concomitant:

* Prior use of any systemic anti-cancer chemotherapy for HCC
* Prior use of systemic investigational agents for HCC
* Prior use of Raf-kinase inhibitors (RKI), VEGF inhibitors, EMK inhibitors or Farnesyl transferase inhibitors
* Major surgery within 4 weeks of start of the study drug
* Use of biologic response modifiers, such as granulocytes colony-stimulating factor (G-CSF) within 3 weeks prior to study entry (G-CSF and other hematopoietic growth factors may be used in the management of acute toxicity such as febrile neutropenia when clinically indicated or at the discretion of the investigator; however they may not be substituted for a required dose reduction)
* Patients taking chronic erythropoietin are permitted provided no dose adjustment is undertaken within 1 month prior to the study or during the study.
* Autologous bone marrow transplant or stem cell rescues within four months of start of study drug
* Concomitant treatment with rifampin and St John's wort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2014-01; Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Overall and disease-free survival genes. | 10 years
  Survival analysis

SECONDARY OUTCOMES:
The predictors of survival ( response to Sorafenib ) | 10 years
  Survival analysis
Potential genetic targets for resistance. | 10 years
  Samples will be sequenced using second generation sequencing comparison between, before and after therapy signature will be identified.

CONTACTS AND LOCATIONS:
Overall Officials: Mazen M Hassanain, MBBS FRCSC PhD, Principal Investigator — King Saud University Medical City, Riyadh,KSA.
Locations (1):
- King Saud University Medical City, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhang BH, Yang BH, Tang ZY. Randomized controlled trial of screening for hepatocellular carcinoma. J Cancer Res Clin Oncol. 2004 Jul;130(7):417-22. doi: 10.1007/s00432-004-0552-0. PMID 15042359
- [Background] Sangiovanni A, Del Ninno E, Fasani P, De Fazio C, Ronchi G, Romeo R, Morabito A, De Franchis R, Colombo M. Increased survival of cirrhotic patients with a hepatocellular carcinoma detected during surveillance. Gastroenterology. 2004 Apr;126(4):1005-14. doi: 10.1053/j.gastro.2003.12.049. PMID 15057740
- [Background] Bruix J, Llovet JM. Major achievements in hepatocellular carcinoma. Lancet. 2009 Feb 21;373(9664):614-6. doi: 10.1016/S0140-6736(09)60381-0. No abstract available. PMID 19231618
- [Background] Livraghi T, Meloni F, Di Stasi M, Rolle E, Solbiati L, Tinelli C, Rossi S. Sustained complete response and complications rates after radiofrequency ablation of very early hepatocellular carcinoma in cirrhosis: Is resection still the treatment of choice? Hepatology. 2008 Jan;47(1):82-9. doi: 10.1002/hep.21933. PMID 18008357
- [Background] Llovet JM, Schwartz M, Mazzaferro V. Resection and liver transplantation for hepatocellular carcinoma. Semin Liver Dis. 2005;25(2):181-200. doi: 10.1055/s-2005-871198. PMID 15918147
- [Background] Thomas MB, O'Beirne JP, Furuse J, Chan AT, Abou-Alfa G, Johnson P. Systemic therapy for hepatocellular carcinoma: cytotoxic chemotherapy, targeted therapy and immunotherapy. Ann Surg Oncol. 2008 Apr;15(4):1008-14. doi: 10.1245/s10434-007-9705-0. Epub 2008 Jan 31. PMID 18236117
- [Background] Mathurin P, Rixe O, Carbonell N, Bernard B, Cluzel P, Bellin MF, Khayat D, Opolon P, Poynard T. Review article: Overview of medical treatments in unresectable hepatocellular carcinoma--an impossible meta-analysis? Aliment Pharmacol Ther. 1998 Feb;12(2):111-26. doi: 10.1046/j.1365-2036.1998.00286.x. PMID 9692685
- [Background] Perilongo G, Maibach R, Shafford E, Brugieres L, Brock P, Morland B, de Camargo B, Zsiros J, Roebuck D, Zimmermann A, Aronson D, Childs M, Widing E, Laithier V, Plaschkes J, Pritchard J, Scopinaro M, MacKinlay G, Czauderna P. Cisplatin versus cisplatin plus doxorubicin for standard-risk hepatoblastoma. N Engl J Med. 2009 Oct 22;361(17):1662-70. doi: 10.1056/NEJMoa0810613. PMID 19846851
- [Background] Liu L, Cao Y, Chen C, Zhang X, McNabola A, Wilkie D, Wilhelm S, Lynch M, Carter C. Sorafenib blocks the RAF/MEK/ERK pathway, inhibits tumor angiogenesis, and induces tumor cell apoptosis in hepatocellular carcinoma model PLC/PRF/5. Cancer Res. 2006 Dec 15;66(24):11851-8. doi: 10.1158/0008-5472.CAN-06-1377. PMID 17178882
- [Background] Adnane L, Trail PA, Taylor I, Wilhelm SM. Sorafenib (BAY 43-9006, Nexavar), a dual-action inhibitor that targets RAF/MEK/ERK pathway in tumor cells and tyrosine kinases VEGFR/PDGFR in tumor vasculature. Methods Enzymol. 2006;407:597-612. doi: 10.1016/S0076-6879(05)07047-3. PMID 16757355
- [Background] McKeage K, Wagstaff AJ. Sorafenib: in advanced renal cancer. Drugs. 2007;67(3):475-83; discussion 484-5. doi: 10.2165/00003495-200767030-00009. PMID 17335301
- [Background] Wilhelm SM, Carter C, Tang L, Wilkie D, McNabola A, Rong H, Chen C, Zhang X, Vincent P, McHugh M, Cao Y, Shujath J, Gawlak S, Eveleigh D, Rowley B, Liu L, Adnane L, Lynch M, Auclair D, Taylor I, Gedrich R, Voznesensky A, Riedl B, Post LE, Bollag G, Trail PA. BAY 43-9006 exhibits broad spectrum oral antitumor activity and targets the RAF/MEK/ERK pathway and receptor tyrosine kinases involved in tumor progression and angiogenesis. Cancer Res. 2004 Oct 1;64(19):7099-109. doi: 10.1158/0008-5472.CAN-04-1443. PMID 15466206
- [Background] Abou-Alfa GK, Schwartz L, Ricci S, Amadori D, Santoro A, Figer A, De Greve J, Douillard JY, Lathia C, Schwartz B, Taylor I, Moscovici M, Saltz LB. Phase II study of sorafenib in patients with advanced hepatocellular carcinoma. J Clin Oncol. 2006 Sep 10;24(26):4293-300. doi: 10.1200/JCO.2005.01.3441. Epub 2006 Aug 14. PMID 16908937